CLINICAL TRIAL: NCT03417895
Title: Anti-PD-1 Antibody SHR-1210 Combined With Anti-angiogenesis Inhibitor Apatinib in Treatment of Extensive-stage Disease Small Cell Lung Cancer After Failure of First Line Standard Therapy
Brief Title: SHR-1210 Combined With Apatinib in Treatment of ED-SCLC After Failure of First Line Standard Therapy
Acronym: PASSION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-II-206
Record Dates: First submitted 2018-01-08; First posted 2018-01-31 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2023-04

CONDITIONS: Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (SHR-1210+Apatinib) (Experimental): SHR-1210 200mg, IV, Q2W and Apatinib 375mg, PO, QD
  Interventions: Drug: SHR-1210; Drug: Apatinib
- B (SHR-1210+Apatinib) (Experimental): SHR-1210 200mg, IV, Q2W and Apatinib 375mg, PO, QD (5 Days on, 2 Days off)
  Interventions: Drug: SHR-1210; Drug: Apatinib
- C (SHR-1210+Apatinib) (Experimental): SHR-1210 200mg, IV, Q2W and Apatinib 375mg, PO, QD (7 Days on, 7 Days off)
  Interventions: Drug: SHR-1210; Drug: Apatinib

INTERVENTIONS:
Drug: SHR-1210 — A humanized anti-PD-1 monoclonal antibody
Drug: Apatinib — A tyrosine kinase inhibitor selectively targeting VEGFR-2

SUMMARY:
This is a multi-center, open-label, phase II study of intravenous (IV) SHR-1210 at 200mg,q2w in combination with Apatinib at one dose (375mg). Comparison of 3 different dose schedules in subjects with extensive-stage disease small cell lung cancer. SHR-1210 is a humanized monoclonal antibody against Programmed death 1(PD-1). Apatinib is a new kind of selective Vascular Endothelial Growth Factor Receptor 2 (VEGFR-2) tyrosine kinase inhibitor (TKI).

The study is composed of two parts. Part 1 of the study will determine the safety and tolerability of SHR-1210 in combination with Apatinib in first 6 subjects of each arm. The second phase of treatment was carried out by selecting one group of administration mode and the tolerated dose of Apatinib. Part 2 of the study will determine the safety and efficacy of SHR-1210 in combination with Apatinib in 39 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Signed inform consent form.
2. Age >= 18 years and <= 70 years.
3. Histologically or cytologically confirmed small cell lung cancer.
4. ED-SCLC according to Veterans Administration Lung Study Group.
5. Radiographically progression following a platinum-based standard prior chemotherapy regimen.
6. Eastern Cooperative Oncology Group performance status of 0 or 1.
7. Measurable disease as defined by RECIST v1.1.
8. Life expectancy >= 8 weeks.
9. Adequate hematologic and end organ function.

Exclusion Criteria:

1. Histologically or cytologically confirmed mixed non-small cell and small cell carcinoma.
2. Prior exposure to therapeutic anticancer vaccines; prior exposure to any T cell co-stimulatory therapy or immune checkpoint inhibitors, including but not limited to other anti-CTLA-4, anti-PD-1, anti-PD-L1 and anti-PD-L2 antibodies.
3. Prior exposure to anti-VEGF or anti-VEGFR therapy.
4. Active brain metastasis or meningeal metastasis.
5. Clinically significant third space effusion (e.g., uncontrolled pericardial effusion, ascites or pleural effusion by extraction or other treatment).
6. Known hypersensitivity to study drug or any of its excipients; known hypersensitivity to any antibody.
7. Treatment with any other investigational agent or participation in another clinical trial within 4 weeks prior to screening.
8. Other conditions that the investigator thinks unsuitable in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Shi, Study Director — Jiangsu Hengrui Pharmaceutical Co., Ltd.
Locations (2):
- China (2):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fan Y, Zhao J, Wang Q, Huang D, Li X, Chen J, Fang Y, Duan J, Zhou C, Hu Y, Yang H, Hu Y, Zhou J, Lin X, Wang L, Wang Z, Xu Y, Zhang T, Shi W, Zou J, Wang J. Camrelizumab Plus Apatinib in Extensive-Stage SCLC (PASSION): A Multicenter, Two-Stage, Phase 2 Trial. J Thorac Oncol. 2021 Feb;16(2):299-309. doi: 10.1016/j.jtho.2020.10.002. Epub 2020 Nov 6. PMID 33166719

RESULTS

PARTICIPANT FLOW:
Groups:
- A(SHR-1210+Apatinib): SHR-1210 200mg, IV, Q2W and Apatinib 375mg, PO, QD
- B(SHR-1210+Apatinib): SHR-1210 200mg, IV, Q2W and Apatinib 375mg, PO, QD (5 Days on, 2 Days off)
- C(SHR-1210+Apatinib): SHR-1210 200mg, IV, Q2W and Apatinib 375mg, PO, QD (7 Days on, 7 Days off)
Period: Overall Study
Arm/Group | A(SHR-1210+Apatinib) | B(SHR-1210+Apatinib) | C(SHR-1210+Apatinib)
Started | 47 | 6 | 6
Completed | 47 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A(SHR-1210+Apatinib) | B(SHR-1210+Apatinib) | C(SHR-1210+Apatinib) | Total
Number analyzed (Participants) | 47 | 6 | 6 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (6.36) | 59.3 (7.39) | 54.2 (10.68) | 59.6 (7.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 0 | 1 | 8
  Male | 40 | 6 | 5 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 47 | 6 | 6 | 59
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 47 | 6 | 6 | 59

OUTCOME MEASURES:

1. Primary Outcome: Adverse Event
Description: Evaluation of adverse event rate according to CTCAE v4.03
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | A(SHR-1210+Apatinib) | B(SHR-1210+Apatinib) | C(SHR-1210+Apatinib)
Number analyzed (Participants) | 47 | 6 | 6
participants | 47 | 6 | 5

2. Primary Outcome: ORR
Description: Objective response rate according to RECIST v1.1 (Response was assessed with CT or MRI using RECIST v1.1, Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to<10 mm; Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Over all response：CR+PR)
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of number of people in FAS
Arm/Group | A(SHR-1210+Apatinib) | B(SHR-1210+Apatinib) | C(SHR-1210+Apatinib)
Number analyzed (Participants) | 47 | 6 | 6
percentage of number of people in FAS | 34.0 [20.9 to 49.3] | 33.3 [4.3 to 77.7] | 33.3 [4.3 to 77.7]

3. Secondary Outcome: OS Rate
Description: Overall survival rate
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of number of people in FAS
Arm/Group | A(SHR-1210+Apatinib) | B(SHR-1210+Apatinib) | C(SHR-1210+Apatinib)
Number analyzed (Participants) | 47 | 6 | 6
percentage of number of people in FAS | 63.8 [48.4 to 75.7] | 66.7 [19.5 to 90.4] | 44.4 [6.6 to 78.5]

4. Secondary Outcome: PFS
Description: Progression-free survival according to RECIST v1.1
Time Frame: Imaging assessment was performed on C1D28 and every 8 weeks after C1D28 until radiographic progressive disease (PD) was documented.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A(SHR-1210+Apatinib) | B(SHR-1210+Apatinib) | C(SHR-1210+Apatinib)
Number analyzed (Participants) | 47 | 6 | 6
months | 3.6 [1.9 to 4.6] | 3.6 [2.7 to 8.3] | 1.2 [0.9 to 19.7]

5. Secondary Outcome: TTR
Description: Time to response according to RECIST v1.1 (Response was assessed with CT or MRI using RECIST v1.1, Time to response (TTR): date of first dose to date of first documented CR or PR)
Time Frame: as for outcome 4
Measure: Median (Full Range); unit: months
Arm/Group | A(SHR-1210+Apatinib) | B(SHR-1210+Apatinib) | C(SHR-1210+Apatinib)
Number analyzed (Participants) | 47 | 6 | 6
months | 1.0 [0.9 to 4.7] | 1.8 [0.9 to 2.7] | 4.6 [0.9 to 8.2]

6. Secondary Outcome: DoR
Description: Duration of response according to RECIST v1.1 (Response was assessed with CT or MRI using RECIST v1.1, Duration of response (DoR): DoR will only be performed in subjects who have a confirmed tumor response (CR or PR) after treatment
Time Frame: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A(SHR-1210+Apatinib) | B(SHR-1210+Apatinib) | C(SHR-1210+Apatinib)
Number analyzed (Participants) | 47 | 6 | 6
months | 6.2 [3.7 to 9.2] | 4.2 [3.6 to 4.7] | 8.0 [4.6 to 11.5]

7. Secondary Outcome: DCR
Description: Disease control rate according to RECIST v1.1 (Response was assessed with CT or MRI using RECIST v1.1; Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to<10 mm; Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Disease control rate (DCR): CR+PR+SD
Time Frame: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of number of people in FAS
Arm/Group | A(SHR-1210+Apatinib) | B(SHR-1210+Apatinib) | C(SHR-1210+Apatinib)
Number analyzed (Participants) | 47 | 6 | 6
percentage of number of people in FAS | 68.1 [52.9 to 80.9] | 100.0 [54.1 to 100.0] | 50.0 [11.8 to 88.2]

8. Secondary Outcome: OS
Description: Overall survival
Time Frame: on average of 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A(SHR-1210+Apatinib) | B(SHR-1210+Apatinib) | C(SHR-1210+Apatinib)
Number analyzed (Participants) | 47 | 6 | 6
months | 8.8 [4.9 to 12.3] | 11.2 [4.9 to NA] — insufficient participants with events | 5.4 [1.5 to NA] — insufficient participants with events

ADVERSE EVENTS:
Time Frame: 24 months
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | A(SHR-1210+Apatinib) | B(SHR-1210+Apatinib) | C(SHR-1210+Apatinib)
All-Cause Mortality (participants affected / at risk) | 17/47 | 1/6 | 2/6
Serious Adverse Events (participants affected / at risk) | 27/47 | 4/6 | 2/6
Other Adverse Events (participants affected / at risk) | 47/47 | 6/6 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A(SHR-1210+Apatinib) (N=47) | B(SHR-1210+Apatinib) (N=6) | C(SHR-1210+Apatinib) (N=6)
Death (General disorders) | 9 | 1 | 0
Progressive disease (General disorders) | 6 | 0 | 1
Pyrexia (General disorders) | 2 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 2 | 0
Platelet count decreased (Investigations) | 4 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Herniated disc (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tumor progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0
Acute heart failure (Cardiac disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A(SHR-1210+Apatinib) (N=47) | B(SHR-1210+Apatinib) (N=6) | C(SHR-1210+Apatinib) (N=6)
Anaemia (Blood and lymphatic system disorders) | 18 | 1 | 0
Lymph node haemorrhage (Blood and lymphatic system disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 3 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 3 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 1 | 0 | 1
Ventricular hypokinesia (Cardiac disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 16 | 2 | 2
Hyperthyroidism (Endocrine disorders) | 2 | 0 | 1
Scleral haemorrhage (Eye disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 14 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 10 | 1 | 2
Constipation (Gastrointestinal disorders) | 10 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 1 | 3
Stomatitis (Gastrointestinal disorders) | 7 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 4 | 2 | 0
Toothache (Gastrointestinal disorders) | 6 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 13 | 3 | 4
Pyrexia (General disorders) | 11 | 0 | 2
Chest discomfort (General disorders) | 4 | 0 | 2
Chest pain (General disorders) | 4 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1
Sluggishness (General disorders) | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 1
Reactive capillary endothelial proliferation (Immune system disorders) | 5 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 28 | 4 | 5
Alanine aminotransferase increased (Investigations) | 22 | 2 | 3
White blood cell count decreased (Investigations) | 20 | 4 | 2
Platelet count decreased (Investigations) | 20 | 3 | 1
Weight decreased (Investigations) | 21 | 1 | 1
Neutrophil count decreased (Investigations) | 14 | 4 | 2
Blood bilirubin increased (Investigations) | 14 | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 8 | 2 | 1
Blood creatinine increased (Investigations) | 6 | 3 | 1
Blood thyroid stimulating hormone increased (Investigations) | 8 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 7 | 2 | 0
Protein urine present (Investigations) | 7 | 2 | 0
Occult blood positive (Investigations) | 4 | 4 | 0
Blood urea increased (Investigations) | 3 | 1 | 1
Tri-iodothyronine decreased (Investigations) | 5 | 0 | 0
Blood bilirubin unconjugated increased (Investigations) | 3 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 3 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 3 | 0 | 1
Haemoglobin decreased (Investigations) | 2 | 1 | 1
Urinary occult blood positive (Investigations) | 3 | 1 | 0
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 1 | 0 | 2
Bilirubin conjugated increased (Investigations) | 3 | 0 | 0
Protein total decreased (Investigations) | 2 | 0 | 1
Thyroxine free decreased (Investigations) | 2 | 1 | 0
Transaminases increased (Investigations) | 2 | 1 | 0
Blood creatine phosphokinase MB increased (Investigations) | 1 | 0 | 1
Electrocardiogram T wave abnormal (Investigations) | 1 | 0 | 1
Lipase increased (Investigations) | 0 | 2 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 1
Blood cholinesterase decreased (Investigations) | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 1
Electrocardiogram T wave amplitude decreased (Investigations) | 0 | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 1
Glucose urine present (Investigations) | 0 | 1 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 18 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 4 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 6 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 1 | 0
Proteinuria (Renal and urinary disorders) | 18 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 2 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 17 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 9 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 28 | 6 | 3
Thrombosis (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All clinical study findings and documents will be regarded as confidential. The investigator and members of his/her research team must not disclose such information without prior written approval from the sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/95/NCT03417895/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT03417895/SAP_001.pdf